CLINICAL TRIAL: NCT02495090
Title: Hypospadias and Exome: Identification of New Genes for Familial Hypospadias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9477; 2014-A01425-42 (Other: ANSM)
Record Dates: First submitted 2015-06-15; First posted 2015-07-13 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hypospadias
Keywords: Hypospadias; exome sequencing; genital malformation
MeSH Terms: conditions — Hypospadias | interventions — Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypospadias (Other): Familial hypospadias trios (patients + parents)
  Interventions: Genetic: Exome sequencing

INTERVENTIONS:
Genetic: Exome sequencing — Plain DNA sequencing

SUMMARY:
Hypospadias is the second most common malformation of the male genitalia and consists in a congenital hypoplasia of its ventral face. Hypospadias results from abnormal development of the penis that leaves the urethral meatus proximal to its normal glanular position. Meatus position may be located anywhere along the penile shaft, but more severe forms of hypospadias may have a urethral meatus located at the scrotum or perineum. Glandular and penile anterior represents approximately 70% of all the diagnosed cases.

The frequency of family reached depend on the severity of hypospadias. The number of children which have hypospadias mutation discovered by classical technique is low. Families are often the cause of the discovery of new genes involved in sexual differentiation because they allow comparison of genomes of related persons, and detect more easily mutations.

DETAILED DESCRIPTION:
The aim of this protocol is to search for new genes involved in genital malformations such as hypospadias. Addressed to families with usual causes of these malformations excluded. The search for these mutations will be done by exome sequencing in families where several cases of hypospadias were identified.

ELIGIBILITY:
Inclusion Criteria:

* Hypospadiac patients with a familial history of hypospadias

Exclusion Criteria:

* Hypospadiac patients without a family history of hypospadias
* Hypospadiac patients with a family history of hypospadias where etiology is identified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2015-11-12 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
number of new genetic variants | 1 day
  exome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Kalfa, MD, PhD, Principal Investigator — UH Montpellier
Locations (1):
- Hôpital Lapeyronie, Montpellier, France